CLINICAL TRIAL: NCT06203782
Title: Comparison of Endoscopic Strictureplasty and Endoscopic Balloon Dilation for the Treatment of Crohn's Disease Intestinal Strictures: An Open-Label, Multicenter, Randomized Controlled Trial
Brief Title: Comparing Endoscopic Strictureplasty vs. Balloon Dilation in Crohn's Disease Strictures
Acronym: ES vs BD in CD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0877
Record Dates: First submitted 2023-09-28; First posted 2024-01-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the experimental group, 51 patients underwent endoscopic stricturoplasty. A transparent cap was mounted on the front end of the endoscope, and a needle knife was inserted through the working channel of the endoscope. Under direct visualization, a radial incision was made at the site of the stricture, with an effort to preserve normal mucosal tissue as much as possible. The stricture was gradually incised until the endoscope could smoothly pass through.
  Interventions: Procedure: endoscopic stricturoplasty
- Control Group (Experimental): In the control group, 51 patients underwent endoscopic balloon dilation. The endoscope was advanced to the site of the stricture, and a dilation guidewire was inserted. After placing the balloon, it was progressively inflated with pressure, each inflation lasting 1-2 minutes, and this process was repeated 2-3 times until the endoscope and sheath could pass through the narrowed segment and enter the distal colon.
  Interventions: Procedure: endoscopic balloon dilation

INTERVENTIONS:
Procedure: endoscopic stricturoplasty — Experimental Group: In the experimental group, 51 patients underwent endoscopic stricturoplasty. A transparent cap was mounted on the front end of the endoscope, and a needle knife was inserted through the working channel of the endoscope. Under direct visualization, a radial incision was made at the site of the stricture, with an effort to preserve normal mucosal tissue as much as possible. The stricture was gradually incised until the endoscope could smoothly pass through.
  Arms: Experimental Group
Procedure: endoscopic balloon dilation — Control Group: In the control group, 51 patients underwent endoscopic balloon dilation. The endoscope was advanced to the site of the stricture, and a dilation guidewire was inserted. After placing the balloon, it was progressively inflated with pressure, each inflation lasting 1-2 minutes, and this process was repeated 2-3 times until the endoscope and sheath could pass through the narrowed segment and enter the distal colon.
  Arms: Control Group

SUMMARY:
Crohn's disease (CD) is an inflammatory bowel disease characterized by chronic ulcers, strictures, and penetrating lesions in the intestinal tract. In the early stages of the disease, inflammation and ulcers are the primary manifestations. However, as the disease progresses and recurs over the years, even with medication treatment, 30%-50% of patients continue to experience varying degrees of intestinal narrowing, with a percentage of it being irreversible fibrotic strictures.

For CD-associated intestinal fibrotic strictures, drug therapy often yields limited results, and long-term use of biologics may potentially induce or worsen intestinal narrowing. In comparison to medical treatment, surgical intervention offers a more definitive solution for intestinal strictures. However, surgical treatment is invasive and comes with risks of postoperative complications and disease recurrence.

Endoscopic therapy serves as a bridge between medical and surgical treatment options. Key techniques of endoscopic therapy include endoscopic balloon dilation (EBD), endoscopic stricturoplasty (EST), and endoscopic stent placement.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD) is a group of chronic, recurrent, nonspecific inflammatory disorders of the gastrointestinal tract, the etiology of which remains unclear. It primarily encompasses Ulcerative Colitis (UC) and Crohn's Disease (CD). In recent years, the incidence of IBD in China has sharply increased alongside industrialization and urbanization trends. Specifically, the incidence of CD in North America ranges from 6.3 to 23.8 per 100,000 individuals per year, while in China, it is approximately 10.04 per 100,000 individuals per year with an annual growth rate of 1.1%. CD is characterized by chronic ulcers, strictures, and transmural lesions, primarily affecting young adults aged 15 to 25, and it often follows a relapsing and unremitting course. Persistent inflammation in CD can lead to local fibrosis, narrowing of the intestinal lumen, resulting in intestinal strictures and ultimately causing obstructions, significantly impacting both societal productivity and individual quality of life.

Intestinal stricture is one of the most common local complications of CD, often occurring in the ileocecal region and postoperative anastomotic sites. Recent epidemiological studies in China have indicated that nearly 30% of CD patients experience intestinal strictures, consistent with data from other Asian countries. Reports show that approximately 20% of CD patients present with intestinal strictures at the time of diagnosis, with about one-third progressing to strictures within ten years of diagnosis. Moreover, up to 50% of patients will undergo at least one surgical intervention, and about one-quarter will experience stricture recurrence within five years after surgery. CD-related intestinal strictures often combine both inflammatory and fibrotic components. Inflammatory strictures result from mucosal congestion, edema, and lymphoid tissue hyperplasia caused by inflammatory responses in the intestinal wall, which can be relieved by controlling inflammation and reducing tissue edema. Fibrotic strictures, on the other hand, are due to the deposition of fibrous tissue and scarring in the intestinal wall resulting from long-term chronic inflammation, leading to luminal narrowing and even occlusion, with current drug therapies unable to reverse fibrosis.

The three main treatment modalities for CD-related intestinal strictures include medical therapy, endoscopic therapy, and surgical intervention. Medical therapy is generally used for the prevention and management of inflammatory strictures but has limited efficacy against fibrotic strictures. Prolonged use of biologics may induce or exacerbate intestinal strictures, and it is ineffective for anastomotic strictures. Compared to medical therapy, surgical treatment, which includes intestinal resection and anastomotic strictureplasty, offers more definitive results in the treatment of intestinal strictures. However, surgery is invasive and carries risks of postoperative complications and disease recurrence.

Endoscopic therapy has emerged as a bridge between medical and surgical treatments and can be employed to control the progression of intestinal strictures with proven efficacy and a lower risk of complications. Key endoscopic techniques include Endoscopic Balloon Dilation (EBD), Endoscopic Stricturectomy (EST), and stent placement. EBD is the most commonly used endoscopic treatment, involving the placement of a balloon dilator under direct endoscopic visualization or with the assistance of a guidewire, for dilating the narrowed luminal tract of the digestive system. Over the past 30 years, EBD has become a routine treatment for primary and secondary intestinal strictures in CD. EBD achieves immediate success as endoscopy can smoothly navigate through the narrowed segment, with clinical improvement primarily measured by relief of obstructive symptoms. Numerous observational clinical studies have indicated that EBD has a good safety profile and an overall success rate ranging from 58.0% to 80.8%. EBD can extend the interval between surgeries for CD patients with ileocolonic anastomotic strictures and is also effective for patients in the progressive phase with a high risk of multiple surgeries. However, during EBD, many cases require repeated dilations, which can increase the risk of perforation. Studies have reported a combined perforation rate of approximately 3%, along with a relatively high stricture recurrence rate. Although most patients can avoid surgery after multiple dilations, some may eventually require surgical treatment.

EST is a novel and minimally invasive therapy for strictures in the gastrointestinal tract, offering advantages such as ease of operation, high safety, small incisions, and low recurrence rates. EST has been successfully used to treat strictures in various locations, including the bile duct, esophagus, and gastrointestinal tract, achieving favorable treatment outcomes. However, EST requires greater technical proficiency. To perform safe and effective endoscopic stricturectomy, endoscopists must master both endoscopy and the cutting device. EST involves cutting the narrowed area of the intestine under endoscopic guidance using an electric knife, allowing targeted treatment of fibrotic segments and avoiding the risk of perforation associated with even balloon pressure distribution. Compared to EBD, EST offers better dilating effects and a lower risk of perforation. It is particularly effective for primary fibrotic strictures or anastomotic strictures. In a study by Lan et al., 11.3% of CD patients who received EST required further surgery, with only 5 adverse events reported. The proportion of CD patients requiring secondary treatment decreased from 33.5% with EBD to 9.5% with EST in a retrospective study. In another retrospective study, 85 IBD patients showed significant improvement in intestinal strictures after EST treatment, with only 13 patients requiring surgical resection during follow-up, along with 10 reported surgical complications. These data indicate that EST is highly effective and safe. The clinical and research significance of determining whether this new, safe, effective, and low-recurrence treatment is suitable for Chinese CD patients with strictures, and whether it offers advantages over EBD, is of paramount importance.

Although EST technology has shown promise in the treatment of gastrointestinal strictures, its role in CD-related strictures requires further clarification. Currently, there is no comparative study between EST and EBD. Therefore, this project proposes to design a randomized controlled trial comparing EST and EBD for the treatment of CD-related strictures, utilizing a randomized parallel control design to compare the treatment outcomes, complications, and recurrence rates of CD patients undergoing EST or EBD. This study aims to deeply analyze and compare the feasibility, efficacy, and safety of EST and EBD in practical applications.

In summary, this project plans to conduct a randomized controlled trial on adult subjects with CD-related strictures treated with EST or EBD. It will employ techniques such as endoscopy, gastrointestinal imaging, and inflammatory marker monitoring to investigate the clinical remission effects, complications, and recurrence rates of this novel endoscopic treatment on CD patients in China. The study will lay the foundation for further multicenter research with larger sample sizes and provide a new approach for developing CD-related stricture treatment options with higher patient compliance. The successful implementation of this project will reveal the application value and prospects of EST in the treatment of CD-related strictures, offering a reliable treatment option for CD patients and improving their disease symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 75 years old. Clear evidence of primary or secondary strictures in Crohn's disease that can be identified through imaging and endoscopy (colonoscopy can reach the site).

If the patient has previously undergone endoscopic treatment, they must have remained asymptomatic for at least one year.

Complete or partial intestinal obstruction. Ineffectiveness of traditional and step-up treatment approaches. Stricture length less than 5 cm. A maximum of two strictures. Signed informed consent.

Exclusion Criteria:

Strictures complicated by abscesses, fistulas, or other active lesions that are not confined to the stricture site.

Strictures that have previously been treated with stents or dilation, but without symptomatic relief maintained for more than one year.

Pregnancy or lactation. Inability to undergo endoscopic treatment. Severe coagulation disorders (platelet count less than 70,000, INR greater than 1.5).

Concurrent advanced-stage tumors or other severe systemic comorbidities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Remission rate of patients | 1 year
  Number of patients who did not require new endoscopic or surgical treatment due to symptom recurrence within one year of follow-up, quantified and reported.

SECONDARY OUTCOMES:
Safety of both treatment modalities | 1 year
  Incidence and severity of adverse events (including bleeding, perforation, etc.) associated with each treatment modality, as assessed and classified according to standard medical guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Chen, phd, Study Chair — Department of Gastroenterology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 浙江大学医学院第二附属医院, Hangzhou, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
The result of questionnaire can be shared
Supporting Information: Study Protocol
Time Frame: now is available
Access Criteria: All the doctors